CLINICAL TRIAL: NCT05556785
Title: Association of Epicardial Adipose Tissue Volume Axnd Radiodensity With Coronary Artery Calcification in Patients With HFpEF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dongying Zhang, Clinical Professor, Chongqing Medical University
Other Study IDs: DZhang
Record Dates: First submitted 2022-09-23; First posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Heart Failure With Preserved Ejection Fraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Recruiting patients who were diagnosed with HFpEF. Using Non-contrast CT to measure the total Agatston coronary artery calcification score, epicardial adipose tissue volume and attenuation. Analysing the correlation between them.

DETAILED DESCRIPTION:
The study enrolled patients who were diagnosed with HFpEF and admitted to the Cardiology Department of the First Affiliated Hospital of Chongqing Medical University. Using Non-contrast CT to measure the total Agatston coronary artery calcification score, epicardial adipose tissue volume and attenuation. Finally, analysing the correlation between them.

ELIGIBILITY:
Inclusion Criteria:

* Typical symptoms and signs of heart failure
* Left ventricular ejection fraction≥50%
* HFA-PEFF score≥5

Exclusion Criteria:

* severe myocarditis, malignant tumors, liver or renal insufficiency, severe valvular heart disease, and received a bypass surgery or other open-heart surgery

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were diagnosed with HFpEF and admitted to the Cardiology Department of the First Affiliated Hospital of Chongqing Medical University.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Association of epicardial adipose tissue volume axnd radiodensity with coronary artery calcification in Patients with HFpEF | 2022.09
  Using SPSS software to analysis the relationship of epicardial adipose tissue volume axnd radiodensity with coronary artery calcification in Patients with HFpEF

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, China